CLINICAL TRIAL: NCT04644445
Title: Impact of High-Protein Bariatric Diet on the Prevention of Postoperative Nausea and Vomiting
Brief Title: Prevention of Postoperative Nausea and Vomiting After Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 20D.841
Record Dates: First submitted 2020-11-02; First posted 2020-11-25 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Bariatric Surgery Candidate; Postoperative Nausea and Vomiting; Morbid Obesity
Keywords: Bariatric Surgery; Sleeve Gastrectomy; Postoperative Diet; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard bariatric clear liquid diet to be started 4 hours after surgery
- Intervention (Experimental): Bariatric full liquid diet (clear liquid diet + protein shakes) to be started 4 hours after surgery
  Interventions: Dietary Supplement: Bariatric Full Liquid Diet

INTERVENTIONS:
Dietary Supplement: Bariatric Full Liquid Diet — Patient's will receive a Bariatric Full Liquid Diet (standard bariatric clear liquid diet + protein shakes) to be started 4 hours after surgery
  Arms: Intervention

SUMMARY:
Postoperative nausea and vomiting are common occurrences following bariatric surgery, occurring in up to 80% of patients and contributing to increased healthcare utilization and delays in discharge. This study aims to evaluate the impact of a high-protein liquid diet on postoperative nausea, vomiting, and length of stay after laparoscopic or robotic sleeve gastrectomy.

DETAILED DESCRIPTION:
Patients with obesity or morbid obesity who are scheduled to undergoing robotic or laparoscopic sleeve gastrectomy will be screened at their preoperative visit. If they meet inclusion/exclusion criteria, they will be invited to participate in the study and written informed consent will be obtained. If the patient consents to participation, they will be randomized to either the control arm or intervention arm. All patients will undergo sleeve gastrectomy in a standard fashion, either laparoscopically or robotically, as discussed with their bariatric surgeon. Post-operative diet will be initiated 4 hours after surgery. The specific diet received will depend on which arm the patient is randomized into. Post-operative assessments will be completed at various time points for all patients. These include a Verbal Rating Scale of Nausea and Vomiting, Rhodes Index Survey, and Quality of Recover-15 Survey. All patients will track their oral intake on a spreadsheet which will be provided. Additional demographic and clinical data will be collected from the Electronic Medical Record. After hospital discharge, patients will follow up in the clinic one week and one month after surgery, per routine. After the one-month visit, the patient's study participation will be considered complete.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient undergoing robotic or laparoscopic sleeve gastrectomy
* Patient able to provide written informed consent
* Patient able to understand and comply with study guidelines

Exclusion Criteria:

* Inability to provide consent
* Previous history of bariatric or gastroesophageal surgery
* Chronic nausea/vomiting
* Hemoglobin A1C 9 or higher
* Therapeutic anticoagulation
* Celiac disease or gluten sensitivity/intolerance/allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting related delay in hospital discharge | through hospital discharge, an average of two days after surgery
  Inability to be discharged from the hospital on postoperative day 1 due to postoperative nausea and vomiting. This will be measured by inability to maintain oral intake of 4-6 ounces an hour due to feeling of nausea or vomiting.

SECONDARY OUTCOMES:
Length of Stay | through hospital discharge, an average of two days after surgery
  Time from end of surgery to discharge from hospital
Severity of Postoperative Nausea and Vomiting | Baseline until 1 month after surgery
  Patient reported severity based on surveys
Patient Self-Reported Quality of Recovery | Baseline until 1 month after surgery
  Patient reported quality of recovery based on survey
Hospital Antiemetic Usage | through hospital discharge, an average of two days after surgery
  Total amount and type of antiemetic medication received while in the hospital
Cost of Hospital Stay | Up to 30 days after surgery
  Total cost of hospital stay after surgery (including initial admission and any readmissions, ED visits, if applicable)
Weight Loss | Up to 30 days after surgery
  Percent excess weight loss (EWL) and total weight loss (TWL) 1 week and 1 month after surgery
30-Day Events | Up to 30 days after surgery
  Complications, ED Visits, Readmissions

CONTACTS AND LOCATIONS:
Overall Officials: Talar Tatarian, MD, Principal Investigator — Jefferson Health
Locations (2):
- United States (2):
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Methodist Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No